CLINICAL TRIAL: NCT02908763
Title: HBsAg Loss/Seroconversion in Low Replicative Chronic HBV Infection Patients With Low Level HBsAg Treated With Peginterferon Alpha
Brief Title: HBsAg Loss/Seroconversion in Low Replicative Chronic Hepatitis B Virus(HBV) Infection Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Collaborators: Peking University (Other); Huazhong University of Science and Technology (Other); Nanchang University (Other); Huizhou Municipal Central Hospital (Other); First People's Hospital, Shunde China (Other); Shenzhen Third People's Hospital (Other); First People's Hospital of Foshan (Other); Tang-Du Hospital (Other); First Affiliated Hospital of Kunming Medical University (Other); Yuebei People's Hospital (Other)
Responsible Party: Principal Investigator, Zhiliang Gao, chief director of department of infectious disease, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3rd-SYSU-I-Cure-4
Record Dates: First submitted 2016-08-27; First posted 2016-09-21 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Chronic Hepatitis B
Keywords: Chronic Hepatitis B; Peginterferon Alpha
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a; peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pegylated interferon group (Experimental): Low replicative chronic HBV infection patients with HBsAg <1000 IU/ mL and HBV DNA<2000 IU/mL are to receive peginterferon alfa-2a 180 micrograms/week or peginterferon alfa-2b 80 micrograms/week for at most 96 weeks.
  Interventions: Drug: peginterferon alfa
- Observing Group (No Intervention): Only observing and following up in this group.

INTERVENTIONS:
Drug: peginterferon alfa — peginterferon alfa-2a 180 micrograms/week or peginterferon alfa-2b 80 micrograms/week, for at most 96 weeks.
  Other Names: peginterferon alfa-2a or peginterferon alfa-2b
  Arms: Pegylated interferon group

SUMMARY:
HBsAg Loss/Seroconversion is uncommon in Low replicative chronic HBV infection patients. The purpose of this study is to investigate the ability of peginterferon alpha to achieve HBsAg loss/seroconversion therapy in Low replicative chronic HBV infection patients with Low Level HBsAg.

DETAILED DESCRIPTION:
Low replicative chronic HBV infection patients with low Level HBsAg were enrolled in the out-patient department of 3rd Affiliated Hospital of Sun Yat-sen University. All of them were HBsAg positive and anti-HBs negative for more than 6 months with HBV DNA<2000 IU/mL and HBsAg levels ≤1000 IU/mL. All patients did not have other liver diseases and contraindications for interferon therapy.

After giving informed consent, patients were treated with weekly subcutaneous injections of alfa-2a 180 micrograms/week or peginterferon alfa-2b 80 micrograms/week. The use of other immune suppressive or regulatory drugs and other antiviral drugs was prohibited during the course of the study.

In this study, treatment endpoint was HBsAg loss(<0.05 IU/mL) and anti-HBs positive(>10 milli-International unit(mIU)/mL) defined as seroconversion. Depending on the decline of HBsAg level, treatment was either continued for a prolonged period (no more than 96 weeks) until the endpoint was achieved, or terminated in case of nonresponse. Treatment was proceeded if HBsAg level continued to decline until HBsAg seroconversion was achieved and the anti-HBs level was above 200 mIU/ml. If the patients were not willing to extend treatment, the therapy was ended at the time of HBsAg loss, or stopped without further decline of HBsAg levels.

ELIGIBILITY:
Inclusion Criteria:

1. Hepatitis B surface antigen (HBsAg) positive and <1000 IU/mL.
2. Hepatitis B surface antibody (HBsAb) negative.
3. Hepatitis B e antigen (HBeAg) negative.
4. Hepatitis B virus DNA <2000 IU/mL.
5. Absence of previous antiviral therapy.

Exclusion Criteria:

1. Patients with active alcohol and/or drugs consumption.
2. Patients with liver cirrhosis, Hepatocellular Carcinoma or other malignancies.
3. Patients with other factors causing liver diseases.
4. Pregnant and lactating women.
5. Patients with concomitant HIV infection or congenital immune deficiency diseases.
6. Patients with diabetes, autoimmune diseases.
7. Patients with important organ dysfunctions.
8. Patients with mental illness.
9. Patients who receive antineoplastic or immunomodulatory therapy in the past 12 months.
10. Patients who can't come back to clinic for follow-up on schedule.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
HBsAg Clearance Rate | 96 weeks
  Percentage of Participants with HBsAg negative.

SECONDARY OUTCOMES:
HBsAg Seroconversion Rate | 96 weeks
  Percentage of Participants with HBsAg negative and anti-HBsAg positive

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Infectious Diseases, The Third Affliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided